CLINICAL TRIAL: NCT00743782
Title: Comparing Pump vs. Subcutaneous Injection Delivery of PTH 1-34 in the Management of Chronic Hypoparathyroidism
Brief Title: Comparing Pump With Subcutaneous Injection Delivery of PTH 1-34 in the Management of Chronic Hypoparathyroidism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 080203; 08-CH-0203
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Hypoparathyroidism; Hypocalcemia
Keywords: Hypoparathyroidism; Parathyroid Hormone 1-34
MeSH Terms: conditions — Hypoparathyroidism; Hypocalcemia

INTERVENTIONS:
Drug: Synthetic Human Parathyroid Hormone 1-34

SUMMARY:
This study will evaluate the safety, biological activity, and pharmacokinetics of PTH delivered by subcutaneous injection compared with an infusion pump. We anticipate pump delivery of PTH will be more physiologic because it mimics normal parathyroid gland secretion of PTH. We expect that pump delivery will simultaneously normalize blood and urine calcium, phosphorus and magnesium levels with minimal or no fluctuations throughout the day. Pump therapy will require lower PTH doses and should normalize markers of bone turnover. We expect the improved metabolic control during pump therapy will be especially evident in patients with more severe forms of hypoparathyrodism where there is an unmet need for improved therapy.

DETAILED DESCRIPTION:
Prior studies (92-CH-0011) have been important in establishing synthetic human parathyroid hormone 1-34 (PTH) as a beneficial treatment for hypoparathyroidism, superior to conventional therapy with calcium and calcitriol. We are conducting a randomized crossover study comparing twice-daily subcutaneous injections vs. PTH pump therapy. We hypothesize that pump delivery of PTH 1-34, compared to twice-daily administration, will provide smoother metabolic control of serum mineral levels and normalization of urine mineral excretion. The two arms will be divided into an inpatient and an outpatient phase. There will be three inpatient admissions, baseline, 3 months, and 6 months. Subjects will be randomized to either pump therapy or to twice daily injections at the beginning of the study and will cross over to the alternate PTH delivery system (injections vs. pump) at the conclusion of the initial 3-month treatment period.

Patients between 10 and 70 years of age who have had chronic hypoparathyroidism for at least 1 year may be eligible for this study. Participants have two 10- 12-day hospital admissions and one 5-day admission. The first two inpatient admissions are separated by 3-month outpatient periods. Outpatient monitoring will require weekly blood tests and monthly urine tests to monitor mineral levels. After third hospital admission, patients will be placed on conventional therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:

This study will include patients of both genders (ages 7-70) with biochemically confirmed chronic hypoparathyroidism of at least one year duration. Twenty-four subjects will be enrolled.

EXCLUSION CRITERIA:

Subjects who meet any of the following criteria are not eligible for the study:

* Pregnancy
* Patients who are calcium infusion dependent and/or do not respond to calcitriol therapy to maintain normal levels of serum calcium will be excluded.
* Seizure disorder requiring antiepileptic medications.

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-08-22; Primary Completion 2014-04-07 (Actual); Study Completion 2014-04-07 (Actual)

PRIMARY OUTCOMES:
Assess the feasability of PTH 1-34 therapy via pump.

SECONDARY OUTCOMES:
This pilot study is being conducted to compare PTH therapy via pump vs. twice daily subcutaneous injections.

CONTACTS AND LOCATIONS:
Overall Officials: Karen K Winer, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Winer KK, Sinaii N, Peterson D, Sainz B Jr, Cutler GB Jr. Effects of once versus twice-daily parathyroid hormone 1-34 therapy in children with hypoparathyroidism. J Clin Endocrinol Metab. 2008 Sep;93(9):3389-95. doi: 10.1210/jc.2007-2552. Epub 2008 May 20. PMID 18492754
- [Background] Winer KK, Ko CW, Reynolds JC, Dowdy K, Keil M, Peterson D, Gerber LH, McGarvey C, Cutler GB Jr. Long-term treatment of hypoparathyroidism: a randomized controlled study comparing parathyroid hormone-(1-34) versus calcitriol and calcium. J Clin Endocrinol Metab. 2003 Sep;88(9):4214-20. doi: 10.1210/jc.2002-021736. PMID 12970289
- [Background] Winer KK, Yanovski JA, Cutler GB Jr. Synthetic human parathyroid hormone 1-34 vs calcitriol and calcium in the treatment of hypoparathyroidism. JAMA. 1996 Aug 28;276(8):631-6. PMID 8773636
- [Background] Winer KK, Sinaii N, Reynolds J, Peterson D, Dowdy K, Cutler GB Jr. Long-term treatment of 12 children with chronic hypoparathyroidism: a randomized trial comparing synthetic human parathyroid hormone 1-34 versus calcitriol and calcium. J Clin Endocrinol Metab. 2010 Jun;95(6):2680-8. doi: 10.1210/jc.2009-2464. Epub 2010 Apr 14. PMID 20392870
- [Derived] Winer KK, Fulton KA, Albert PS, Cutler GB Jr. Effects of pump versus twice-daily injection delivery of synthetic parathyroid hormone 1-34 in children with severe congenital hypoparathyroidism. J Pediatr. 2014 Sep;165(3):556-63.e1. doi: 10.1016/j.jpeds.2014.04.060. Epub 2014 Jun 16. PMID 24948345